CLINICAL TRIAL: NCT07365852
Title: Accuracy Assessment of Symphyseal Onlay Bone Grafting for 3D Maxillary Ridge Augmentation Using Tooth-supported Patient-specific Surgical Guide Versus Free Hand Technique: A Randomized Controlled Trial
Brief Title: Accuracy Assessment of Chin Graft for Ridge Augmentation Using Tooth-supported Guide Versus Free Hand Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wesam Sami Hassan Ali, Resident at oral and maxillofacial surgery department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4596
Record Dates: First submitted 2024-06-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alveolar Bone Loss
Keywords: ridge augmentation; onlay grafting; tooth-supported guide; patient-specific guide; maxillary bone augmentation; chin graft
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth-supported Patient-specific Surgical Guide (Experimental): In this study computer-designed patient-specific surgical osteotomy guide provides accurate harvesting of autogenous bone blocks from chin area.Then, graft placement will be done using patient-specific tooth-supported guide in upper anterior deficient ridge and fixation using 2 micro screws labially and one through and through for the palatal shell.
  Interventions: Procedure: 3D ridge augmentation using tooth-supported patient-specific guide
- Free hand technique (Active Comparator): The cortical bone harvested from chin area without surgical guide, then the non-guided mono-cortical bone block grafting will be fixed on the ridge labially using 2 micro screws and one through and through for the palatal shell.
  Interventions: Procedure: 3D ridge augmentation using tooth-supported patient-specific guide

INTERVENTIONS:
Procedure: 3D ridge augmentation using tooth-supported patient-specific guide — In this study computer-designed patient-specific surgical osteotomy guide should provide accurate harvesting of autogenous bone blocks from chin area.Then, graft placement will be done using patient-specific tooth-supported guide in upper anterior deficient ridge and fixation using 2 micro screws labially and one through and through for the palatal shell.

SUMMARY:
This study compares the accuracy of osteotomies positions using patient specific guides for onlay bone shells harvested from the chin then the graft positioning for 3D upper anterior ridge augmentation using patient-specific tooth-supported guide versus free hand technique

DETAILED DESCRIPTION:
In this study the tooth-supported stereolithographic guiding template is proposed to allow accurate onlay grafting of labial and palatal mono-cortical shells simultaneously after harvesting using computer-designed patient-specific surgical osteotomy guide. This customized osteotomy guide should provide accurate harvesting of autogenous bone blocks from chin area which also provides suitable contour with the anterior ridge area. This computer assisted surgery is supposed to help in decreasing the operation time, thus decreasing the devascularization time to the bone graft. Thus, it helps for increased accuracy to increase three-dimensional bone gain and decrease morbidity of donor site while gaining the maximum available bone volume. Tooth-supported graft placement guide provides reproducible and convenient design without the need of high surgical skills as well.

ELIGIBILITY:
Inclusion Criteria:

* • Anterior maxilla with horizontal deficient alveolar ridge that is from 2 to 4 mm measured from the crest of the alveolar ridge buccolingually, combined with vertical deficiency.

  * Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
  * Both genders males and females will be included
  * Normal vertical dimension with normal inter-arch space

Exclusion Criteria:

* Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.
* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing females.
* Immunosuppressed or immunocompromised
* Heavy smokers
* Patients undergo medication interfere with bone healing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Alveolar ridge width bone gain | 4 months
  measures will be obtained from CT scan in millimetres

SECONDARY OUTCOMES:
Alveolar ridge vertical bone gain | 4 months
  measures will be obtained from CT scan in millimetres

OTHER OUTCOMES:
Accuracy of the Computer-assisted guide in the study group | immediate post-operative
  measures will be obtained from CT scan in millimetres

CONTACTS AND LOCATIONS:
Overall Officials: Wesam Sami, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aloy-Prosper A, Carramolino-Cuellar E, Penarrocha-Oltra D, Soto-Penaloza D, Penarrocha-Diago M. Intraoral onlay block bone grafts versus cortical tenting technique on alveolar ridge augmentations: a systematic review. Med Oral Patol Oral Cir Bucal. 2022 Mar 1;27(2):e181-e190. doi: 10.4317/medoral.25169. PMID 35218647
- [Background] Cansiz E, Haq J, Manisali M, Cakarer S, Gultekin BA. Long-term evaluation of three-dimensional volumetric changes of augmented severely atrophic maxilla by anterior iliac crest bone grafting. J Stomatol Oral Maxillofac Surg. 2020 Dec;121(6):665-671. doi: 10.1016/j.jormas.2019.11.004. Epub 2020 Feb 8. PMID 32045687
- [Background] Chen ST, Beagle J, Jensen SS, Chiapasco M, Darby I. Consensus statements and recommended clinical procedures regarding surgical techniques. Int J Oral Maxillofac Implants. 2009;24 Suppl:272-8. No abstract available. PMID 19885450
- [Background] De Stavola L, Fincato A, Bressan E, Gobbato L. Results of Computer-Guided Bone Block Harvesting from the Mandible: A Case Series. Int J Periodontics Restorative Dent. 2017 Jan/Feb;37(1):e111-e119. doi: 10.11607/prd.2721. PMID 27977816
- [Background] Naishlos S, Zenziper E, Zelikman H, Nissan J, Mizrahi S, Chaushu G, Matalon S, Chaushu L. Esthetic Assessment Succeeding Anterior Atrophic Maxilla Augmentation with Cancellous Bone-Block Allograft and Late Restoration Loading. J Clin Med. 2021 Oct 9;10(20):4635. doi: 10.3390/jcm10204635. PMID 34682757